CLINICAL TRIAL: NCT01380418
Title: Factors Associated With Chronic Respiratory Failure in Obesity: A Cross-sectional Study
Brief Title: Factors Associated With Chronic Respiratory Failure in Obesity
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Ari Manuel, Ari Manuel, Oxford University Hospitals NHS Trust
Other Study IDs: 11/H0605/9; NCT01385462 (obsolete NCT alias)
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Obesity Hypoventilation Syndrome
Keywords: Obesity
MeSH Terms: conditions — Obesity; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, fat, muscle
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Obese BMI>30 18-85 years old

SUMMARY:
Some overweight individuals develop problems with their breathing such that they gradually breathe less and less. This leads to a lack of oxygen and a buildup of carbon dioxide in the blood, called ventilatory failure. As a consequence, if such a person develops a chest infection, they are more likely to become seriously ill and need intensive care. In addition they are much more likely to develop severe complications during and following operations. This problem can be treated with a machine at home used overnight to help breathing. It is interesting that ventilatory failure only happens in some overweight individuals, and the investigators do not understand what factors make this complication develop. There are a number of theories: for example the distribution of the fat, additional lung disease (such as asthma), the addition of obstructive sleep apnoea, a condition when there are periods of cessation of breathing overnight (which is more common in obese individuals), weak muscles of breathing (perhaps due to fatty infiltration of muscles or vitamin D deficiency), and other hormonal changes.

The investigators intend to measure many potential factors in a range of overweight individuals, some who have ventilatory failure, and some who do not, to try and work out which are the important factors that cause this problem. If the investigators can identify such factors, then this will help predict in advance who is at risk from chest infections and during operations; thus allowing for earlier provision of an overnight breathing machine. This should reduce complications and potentially deaths in such individuals.

DETAILED DESCRIPTION:
To test the hypothesis that in obese patients with obesity-hypoventilation (OHS) there are specific factors related to the development of ventilatory failure, compared to obese subjects not in ventilatory failure

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI > 30) with or without obesity hypoventilation
* (OHS) (18 - 85yrs)
* Admitted for management of their OHS
* Attending the sleep and ventilation clinic
* Being assessed for bariatric surgery
* Willing and able to give informed consent for participation in the study
* Men and women aged 18 - 85 years

Exclusion Criteria:

* Respiratory acidosis pH <7.30
* Severe untreated hypothyroidism
* Current treatment with theophylline
* Current treatment with diuretics
* Severe restrictive or obstructive lung disease (<30% predicted)
* Severe comorbidities such as moderate/severe COPD, left sided heart failure, and primary CNS or neuromuscular diseases
* Contraindications to MRI scanning
* Contraindications to DXA scanning
* Previous participant in research in the last 12 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese (BMI > 30kg/m2) with or without OHS (18-85yrs)
  1. Admitted for management of OHS
  2. Attending the sleep and ventilation clinic
  3. Being assessed for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To determine the physiological between obese patients with OHS and obese patients without OHS | 1 year
  This will be a detailed ventilatory drive measurements and muscle strength testing. The comparison will be made within the group amongst the range of ventilatory failure

CONTACTS AND LOCATIONS:
Overall Officials: John Stradling, FRCP MBBS PHD, Study Director — University of Oxford
Locations (1):
- Oxford Radcliffe NHS Trust Hospitals, Oxford, United Kingdom

REFERENCES:
- [Derived] Dattani RS, Swerner CB, Stradling JR, Manuel AR. Exploratory study into the effect of abdominal mass loading on airways resistance and ventilatory failure. BMJ Open Respir Res. 2016 Jun 9;3(1):e000138. doi: 10.1136/bmjresp-2016-000138. eCollection 2016. PMID 27335651
- [Derived] Manuel AR, Hart N, Stradling JR. Correlates of obesity-related chronic ventilatory failure. BMJ Open Respir Res. 2016 Feb 18;3(1):e000110. doi: 10.1136/bmjresp-2015-000110. eCollection 2016. PMID 26918192
- [Derived] Manuel ARG, Hart N, Stradling JR. Is a raised bicarbonate, without hypercapnia, part of the physiologic spectrum of obesity-related hypoventilation? Chest. 2015 Feb;147(2):362-368. doi: 10.1378/chest.14-1279. PMID 25080050